CLINICAL TRIAL: NCT06917456
Title: The Codesign and Evaluation of a Novel Virtual Reality Intervention for Use in Psychiatric Inpatient Wards
Brief Title: Novel VR Intervention for Use in Psychiatric Inpatient Wards
Status: Recruiting | Type: Observational
Sponsor: South West London and St George's Mental Health NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: OBRA1004
Record Dates: First submitted 2025-03-18; First posted 2025-04-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Mental Health; Virtual Reality
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants from inpatient wards: This cohort will include patients and staff from inpatient psychiatric wards.
  Interventions: Device: Virtual Reality Headset

INTERVENTIONS:
Device: Virtual Reality Headset — Participants will use either a Meta Quest VR device, or a Pico headset. Both of these devices are standard non-medical hardware items.

SUMMARY:
The current study aims to examine the feasibility and acceptability of a VR app for use on inpatient psychiatric wards. The study will be completed in two stages.

Stage One is a co-design stage. A virtual reality hypnotherapy app that has been developed in collaboration with the company Phase Space, will be trialled with psychiatric inpatients. 16 patients and six staff members will be recruited at this stage. The first eight patients will test the headset and provide feedback. Based on this, the app will be modified by Phase Space and then trialled by an additional eight patients. Concurrently with the recruitment of the 16 patients, six staff members from the ward will be recruited to complete an interview about the feasibility and use of virtual reality headsets on the ward. The total feedback will be taken back to Phase Space who will further modify the app to then be implemented in the pilot stage.

Stage Two- Pilot stage. The Pilot stage will be held in the sensory rooms of two inpatient psychiatric wards. The recruitment period will last four weeks. During the four-week period, participants will have the option of attending a drop-in session held on their ward. The drop-in session will be held twice weekly for the four-week period and participants will be able to use the VR headset during this time period. They will be able to attend the drop-in session as frequently as they would like over the four week period, meaning that they have the ability to attend up to eight drop-in sessions. The new app will be piloted on sixteen inpatients to see if it is deemed acceptable and feasible for use on inpatient wards. the first use of the headset, as well as after four sessions (or earlier if the participant decides to end involvement before they reach four sessions). If a participant attends all eight sessions, they will complete the questionnaires again after the eighth session. Additionally, participants will complete the CR Comment Card before and after each use of the VR headset. Participants will also complete a short qualitative interview after their last session. The interview will comprise of asking participants to provide any feedback they have on the VR, as well as understanding more about how they could see the VR implemented into a ward setting.

Staff members will be recruited to assist in the running of the VR drop-in sessions. Staff will also be asked to provide any feedback on the sessions and observations of the sessions through a diary. At the end of the recruitment window, staff will also be asked to complete a short interview asking about topics such as any changes in participants' behaviour after the VR, logistical challenges around patients using the headsets, how the equipment was looked after and maintained, locations used for the VR and demands on staff time for the rollout.

ELIGIBILITY:
Inclusion Criteria:

* Current inpatient or staff member on an inpatient psychiatric ward
* Capacity to consent

Exclusion Criteria:

* Lacking capacity to provide consent
* History of seizures
* Has a pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population in the study will include inpatients and staff from psychiatric inpatient wards.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the virtual reality software | through study completion, an average of 1 month
  Acceptability of the virtual reality software will be measured through the feedback provided in the qualitative interviews with the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Aileen O'Brien, Principal Investigator — South West London & St. George's Mental Health NHS Trust
Locations (1):
- Springfield University Hospital, South West London & St. George's Mental Health NHS Trust, London, United Kingdom